CLINICAL TRIAL: NCT00329095
Title: An Evaluation of Use of Topical Ocular Hypotensive Medication by Electronic Compliance Measures
Brief Title: An Evaluation of Use of Topical Ocular Hypotensive Medication by Compliance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Robin, Alan L., M.D. (Individual)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GMED-01
Record Dates: First submitted 2006-05-19; First posted 2006-05-24 (Estimated); Last update posted 2006-05-24 (Estimated); Status verified 2006-05

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Compliance
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Patient Compliance | interventions — Travoprost; Latanoprost; Bimatoprost

INTERVENTIONS:
Drug: travoprost, latanoprost, or bimatoprost
Drug: Additional ocular hypotensive medication

SUMMARY:
This is an open-label study in patients who are currently using either a topical prostaglandin as sole ocular hypotensive medical therapy q.d., or a topical prostaglandin plus an adjunctive topical ocular hypotensive marketed product either q.d., or b.i.d. in the same eye(s). Compliance will be measured over the two months of participation.

DETAILED DESCRIPTION:
This is an open-label study in patients who are currently using either a topical prostaglandin as sole ocular hypotensive medical therapy q.d., or a topical prostaglandin plus an adjunctive topical ocular hypotensive marketed product either q.d., or b.i.d. in the same eye(s). Compliance will be measured over the two months of participation.

ELIGIBILITY:
Inclusion Criteria:

* Currently using one or two topical ocular hypotensive medications

Exclusion Criteria:

* Hypersensitivity to any component of medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-12; Study Completion 2006-04

PRIMARY OUTCOMES:
Compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Alan L. Robin, MD, Principal Investigator — Alan L. Robin, M.D.

REFERENCES:
- [Derived] Robin AL, Novack GD, Covert DW, Crockett RS, Marcic TS. Adherence in glaucoma: objective measurements of once-daily and adjunctive medication use. Am J Ophthalmol. 2007 Oct;144(4):533-40. doi: 10.1016/j.ajo.2007.06.012. Epub 2007 Aug 8. PMID 17686450